CLINICAL TRIAL: NCT06055998
Title: Frequency ,Etiology and Prognostic Factors of Acute Transverse Myelitis in Neurology and Psychiatry Department, Assiut University
Brief Title: Frequency ,Etiology and Prognostic Factors of Acute Transverse Myelitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fouad E Fawaz, Resident Doctor, Assiut University
Other Study IDs: acute transverse myelitis
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Transverse Myelitis
MeSH Terms: conditions — Myelitis, Transverse

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — MRI SPINE

SUMMARY:
To identify the frequency of ATM and its different aetiologies, alongside the different clinical and radiological patterns and prognostic factors .

DETAILED DESCRIPTION:
Acute transverse myelitis (ATM) is an inflammatory condition of the spinal cord, covering the entire cross section and spreading on two or more vertebral segments, without evidence of a compressive lesion.1 This shows clinically as acute or subacute spinal cord dysfunction resulting in paresis, sensory level, and autonomic (bladder, bowel, and sexual) impairment below the level of the lesion.2 ATM is typically classified as either idiopathic ATM where no causative factor found or disease- associated transverse myelitis.3 Disease- associated transverse myelitis results from heterogenous pathophysiologic causes including infectious, parainfectious, paraneoplastic, drug/toxin-induced, systemic autoimmune disorders (SAIDs), Neurosarcoidosis and acquired demyelinating diseases like multiple sclerosis (MS) or neuromyelitis optica (NMO).4 5 6 The annual incidence of ATM ranges from 1.34 to 4.60 cases per million,7 8 but increases to 24.6 cases per million if acquired demyelinating diseases like MS are included.9 TM can occur at any age, although a bimodal peak in incidence occurs in the second and fourth decades of life.7 8 10 This broad differential can overlap with noninflammatory myelopathies and can be very challenging for clinicians to navigate, causing delays in diagnosis or treatment.11 MRI is essential to rule out compressive causes of these neurologic manifestations, such as tumour, epidural abscess, herniated disc, stenosis of the medullary canal or hematoma. It is also used to show the extension of the lesion and for follow-up progress of these lesions after treatment.12 The lack of large-scale and longitudinal studies has hindered the understanding of this complex disorder.

Approximately 33% of patients recover with little to no lasting deficits, 33% have a moderate degree of permanent disability, and 33% are permanently disabled.13 The disease is often a monophasic illness and will only not recur unless it is secondary to a chronic comorbid condition, highlight the need for early and prompt recognition of aetiology. Steroids and immunosuppression are the only potential treatments for ATM at this time, but there is potential for monoclonal antibody drugs that might alter the disease course if an autoinflammatory process was identified. Although individuals affected by ATM show residual neurologic deficits if they have not recovered to normal within 3-6 months, no report has considered earlier factors that might determine the prognosis of the illness. The objective of this study was to determine frequency of ATM and its different etiologies, clinical and radiological patterns, and the different prognostic factors associated in a large tertiary center in the south of Egypt with a goal to improve awareness of ATM to ensure prompt recognition and treatment

ELIGIBILITY:
Inclusion Criteria:

Diagnostic criteria include:

1. Sensory, motor, or autonomic dysfunction originating from the spinal cord
2. T2 hyperintense signal changes on MRI
3. No evidence of a compressive lesion
4. Bilateral signs/symptoms.
5. Clearly defined sensory level.
6. Evidence of inflammatory process demonstrated by gadolinium enhancement on MRI, cerebrospinal fluid (CSF) analysis showing pleocytosis, or elevated immunoglobulin G (IgG) index.
7. Progression to nadir between 4 hours and 21 days.

Exclusion Criteria:

1. An alternative diagnosis became apparent any time along the study period including evidence of compressive lesion in MRI, history of previous radiation to the spine within the past 10 years, clinical deficit consistent with thrombosis of the anterior spinal artery or Abnormal flow voids on the surface of the spinal cord consistent with AVFs.
2. Incomplete clinical, laboratory or radiographic data.
3. Patients refused to sign the informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases of all ages and both sex attending the neurology and psychiatry department at Assiut
  University Hospital during one year period who meet the diagnostic criteria of ATM according to the TM
  Consortium Working Group (TMCWG) in 2002 will be recriuted
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Determine the relative frequency of different aetiologies of ATM among Southern Egyptian patients attending Assiut University Hospital | 1 year
  All cases of all ages and both sex attending the neurology and psychiatry department at Assiut University Hospital during one year period who meet the diagnostic criteria of ATM according to the TM
  Consortium Working Group (TMCWG) in 2002 will be recriuted.1 Diagnostic criteria include:
  1. Sensory, motor, or autonomic dysfunction originating from the spinal cord
  2. T2 hyperintense signal changes on MRI
  3. No evidence of a compressive lesion
  4. Bilateral signs/symptoms.
  5. Clearly defined sensory level.
  6. Evidence of inflammatory process demonstrated by gadolinium enhancement on MRI, cerebrospinal fluid (CSF) analysis showing pleocytosis, or elevated immunoglobulin G (IgG) index.
  7. Progression to nadir between 4 hours and 21days.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Youssef, Professor, Study Director — Supervisor; Doaa M Mahmoud, Lecturer, Study Director — Supervisor

REFERENCES:
- [Result] Harizi E, Shemsi K, Kola E, Hyseni F, Kola I, Siddique MA, Sadeque J, Decka A, Dervishi M, Nasir F, Capi L, Ayala I, Ghosh AS, Swarna SS, Musa J, Ahmetgjekaj I. Transverse myelitis in a 26-year-old male with tuberculosis. Radiol Case Rep. 2022 Aug 1;17(10):3669-3673. doi: 10.1016/j.radcr.2022.06.091. eCollection 2022 Oct. PMID 35936885
- [Result] Murthy JM, Reddy JJ, Meena AK, Kaul S. Acute transverse myelitis: MR characteristics. Neurol India. 1999 Dec;47(4):290-3. PMID 10625901
- [Result] Beh SC, Greenberg BM, Frohman T, Frohman EM. Transverse myelitis. Neurol Clin. 2013 Feb;31(1):79-138. doi: 10.1016/j.ncl.2012.09.008. PMID 23186897
- [Result] Christensen PB, Wermuth L, Hinge HH, Bomers K. Clinical course and long-term prognosis of acute transverse myelopathy. Acta Neurol Scand. 1990 May;81(5):431-5. doi: 10.1111/j.1600-0404.1990.tb00990.x. PMID 2375246
- [Result] Bhat A, Naguwa S, Cheema G, Gershwin ME. The epidemiology of transverse myelitis. Autoimmun Rev. 2010 Mar;9(5):A395-9. doi: 10.1016/j.autrev.2009.12.007. Epub 2009 Dec 24. PMID 20035902
- [Result] Debette S, de Seze J, Pruvo JP, Zephir H, Pasquier F, Leys D, Vermersch P. Long-term outcome of acute and subacute myelopathies. J Neurol. 2009 Jun;256(6):980-8. doi: 10.1007/s00415-009-5058-x. Epub 2009 Feb 28. PMID 19252779
- [Result] Berman M, Feldman S, Alter M, Zilber N, Kahana E. Acute transverse myelitis: incidence and etiologic considerations. Neurology. 1981 Aug;31(8):966-71. doi: 10.1212/wnl.31.8.966. PMID 7196523
- [Result] Wingerchuk DM. Postinfectious encephalomyelitis. Curr Neurol Neurosci Rep. 2003 May;3(3):256-64. doi: 10.1007/s11910-003-0086-x. PMID 12691631
- [Result] Jacob A, Weinshenker BG. An approach to the diagnosis of acute transverse myelitis. Semin Neurol. 2008 Feb;28(1):105-20. doi: 10.1055/s-2007-1019132. PMID 18256991
- [Result] de Seze J, Stojkovic T, Breteau G, Lucas C, Michon-Pasturel U, Gauvrit JY, Hachulla E, Mounier-Vehier F, Pruvo JP, Leys D, Destee A, Hatron PY, Vermersch P. Acute myelopathies: Clinical, laboratory and outcome profiles in 79 cases. Brain. 2001 Aug;124(Pt 8):1509-21. doi: 10.1093/brain/124.8.1509. PMID 11459743
- [Result] Frohman EM, Wingerchuk DM. Clinical practice. Transverse myelitis. N Engl J Med. 2010 Aug 5;363(6):564-72. doi: 10.1056/NEJMcp1001112. No abstract available. PMID 20818891
- [Result] Dumic I, Vitorovic D, Spritzer S, Sviggum E, Patel J, Ramanan P. Acute transverse myelitis - A rare clinical manifestation of Lyme neuroborreliosis. IDCases. 2018 Dec 29;15:e00479. doi: 10.1016/j.idcr.2018.e00479. eCollection 2019. PMID 30622896
- [Result] Transverse Myelitis Consortium Working Group. Proposed diagnostic criteria and nosology of acute transverse myelitis. Neurology. 2002 Aug 27;59(4):499-505. doi: 10.1212/wnl.59.4.499. PMID 12236201